CLINICAL TRIAL: NCT05471167
Title: Non-specific Effects of BCG in Under-five Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Inês Fronteira, Assistant professor, Universidade Nova de Lisboa
Other Study IDs: EXPL/SAU-EPI/0067/2021
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Immunity, Heterologous
Keywords: BCG; Mortality; Morbidity; Under 5 children; Immunity, Heterologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Birth cohort 2010: Children born from 01/07/2010 followed up until 30/06/2016
  Interventions: Biological: BCG
- Birth cohort 2011: Children born from 01/07/2011 followed up until 30/06/2017
  Interventions: Biological: BCG
- Birth cohort 2012: Children born from 01/07/2012 followed up until 30/06/2018
  Interventions: Biological: BCG
- Birth cohort 2013: Children born from 01/07/2013 followed up until 30/06/2019
  Interventions: Biological: BCG
- Birth cohort 2014: Children born from 01/07/2014 followed up until 30/06/2020
  Interventions: Biological: BCG
- Birth cohort 2015: Children born from 01/07/2015 followed up until 30/06/2021
  Interventions: Biological: BCG
- Birth cohort 2016: Children born from 01/07/2016 followed up until 30/06/2022
- Birth cohort 2017: Children born from 01/07/2017 followed up until 30/06/2022
- Birth cohort 2018: Children born from 01/07/2018 followed up until 30/06/2022
- Birth cohort 2019: Children born from 01/07/2019 followed up until 30/06/2022
- Birth cohort 2020: Children born from 01/07/2020 followed up until 30/06/2022

INTERVENTIONS:
Biological: BCG — Exposure is defined as having received the BCG vaccine during the first year of life.
  Groups: Birth cohort 2010; Birth cohort 2011; Birth cohort 2012; Birth cohort 2013; Birth cohort 2014; Birth cohort 2015

SUMMARY:
Studies have demonstrated that the reduction in mortality and morbidity due to vaccination extends beyond the targeted infections. This seems to result from the non specific effects of vaccines. BCG, a live attenuated vaccine against TB disease, administered to new borns, is one of the vaccines known to have non specific effects.

In Portugal, between 1965 and June 2016, BCG was administered to all new borns. In July 2016, a clinical guideline established that only children under 6 years of age from high-risk groups should be vaccinated. In 2021, the first cohort of children not vaccinated for BCG reached 5 years of age and evidence is needed on the impact of this strategy.

Aim: to investigate the incidence of specific and non-specific effects of BCG by comparing the incidence of TB disease and infection, mild and severe morbidity, and mortality in the first 5 years of life of children born between 2010 and 2021 according to their BCG status.

Methods: historical birth cohort study of children born between 1st July 2010 and 30th June 2021. The investigators will create a single database that links data from the birth registry, the vaccination registry, the information systems of death certificates, epidemiological surveillance and TB surveillance, Diagnosis Related Groups and of primary health care of children born in the study period to reconstruct chronological sequences of morbidity and mortality events from birth until completion of 5 years of life or 30th June 2021. Only children born in Portugal, live-births and births coded as normal new-born will be included. New borns with low-birth weight (<2kg), premature (<37 weeks) and known or suspected HIV infections will not be included in the study. The follow-up period will be until completion of 5 years of age or 30th June 2022. Data will be analysed to compare the incidence of all-cause mortality (including TB), TB disease and severe and mild morbidity among BCG vaccinated and non-vaccinated children born during the reference period in a total of 11 birth cohorts and will comprise computation of person-time incidence rates for primary outcomes and the probability of surviving (Kaplan Meier method) first and fifth year of life or of not having a hospitalization, emergency department visit or a mild morbidity episode during the follow-up period according to exposure. To explore the effects of several variables on the survival outcomes we will use proportional hazards regression analysis.

DETAILED DESCRIPTION:
Hypothesis: some of the variation observed in child and under-5 mortality, in the incidence of TB, and in severe and mild morbidity in under-5 children might be partially explained by a reduction in coverage rate of BCG since 2016. The reduction in the BCG coverage rate, that resulted from only high-risk children receiving BCG at birth, might have prevented non-vaccinated children from developing trained immunological responses as effectively as BCG vaccinated children.

Aim: to investigate the incidence of specific and non-specific effects of BCG by comparing the incidence of TB disease and infection, mild and severe morbidity and mortality in their first five years of life of children born between 2010 and 2021 according to their BCG status.

Methods Study design: Population based historical (retrospective) birth cohort study Setting : The researchers will investigate the specific and non-specific effects of BCG based on the shift in the BCG vaccination policy that occurred in Portugal in July 2016, when a consistent low incidence of TB led to the revision of the National Immunization Plan. Since then, BCG started to be administered only to new-borns considered to be at higher risk of TB infection, thus creating an opportunity to compare BCG vaccinated and non-vaccinated children.

Participants: Under-5 children born and registered in Portugal between 1 July 2010 and 30 June 2021. This time period will allow to compare the cohorts and exposed and non-exposed to BCG children before and after the 2016 change in the BCG immunization strategy and characterize children not vaccinated with BCG and their health outcomes.

Eligibility criteria: children born in Portugal, live-births and births coded as normal new-born Exclusion criteria: new borns with low-birth weight (<2kg), premature (<37 weeks) and known or suspected HIV infections will not be included in the study.

Follow-up period: until completion of 5 years of age or 30 June 2022. Data sources / measurement: birth registry, vaccination registry, the information systems of death certificates, epidemiological surveillance of notifiable diseases and TB Diagnosis Related Groups and primary health care. These systems contain information on: sex, date of birth, nationality, socioeconomic status, place of residence, health of the mother, health of the new-born (including if BCG was administered at the maternity), and primary health care unit where the child is to be followed up, cause and date of death and date of death, vaccines administrated, date of vaccination, and place of residence, hospitalizations and emergency department visits in public hospitals (including date of admission and discharge, diagnosis and type of admission, motive for admission, weight at birth, DRG code, MDC code), visits to primary health care units and motive, presentation of TB, date of diagnosis, type of treatment, other diseases before TB, risk groups and outcome.

Exposure: having received the BCG vaccine during the first year of life. Measured using the vaccination registry and variables are defined as BCG (Y/N, number of doses) and time from birth to BCG (in days).

Primary outcomes:

Death: death (Y/N); age at time of death (in days); and cause of death. Data on TB diagnosis will include confirmed case (Y/N), presentation of TB, age at diagnosis (in days), duration of treatment and outcome of treatment.

Severe morbidity: hospitalization and visits to the emergency department of the national health system and will include hospital admissions and emergency department visits during the follow-up period (Y/N and number), age (in days) at hospital admission or emergency department visits, length of stay for hospitalizations (in nights); major diagnostic categories for hospitalization and emergency department visits.

Mild morbidity: contacts with the medical doctor or nurse at a primary health centre unit due to disease or ill-health during the follow-up, besides contacts related to recommended child-surveillance scheme or other reasons besides health. Measured through visits to primary health care centre due to disease/ ill-health (Y/N and number), age at visits (in days) and diagnosis.

Mortality and morbidity pertaining to external causes and accidents will not be included in the analysis.

Secondary outcomes: mortality and morbidity profile of under-5 children between 2010 and 2022; the profile of non-vaccinated children before and after 2016, and hospital and primary health care utilization profile of under-5 children.

Statistical methods The researchers will identify, in each database, the data needed and whether a unique identifier exists and can be provided with the dataset. In case a unique identifier is provided, researchers will combine information based on that unique identifier. In case a unique identifier is not provided (most probable scenario) data linkage will be done using a range of proxy identifiers (e.g., date and place of birth, sex, place of residence) to identify probable matches. The type of data linkage method to be used will depend on the type and quality of the linkage variables available on the datasets. However, it is anticipated to have to use a combination of deterministic and probabilistic methods. Before applying linkage methods, data will be cleaned and standardized data, thus identifying and removing errors and inconsistencies (e.g. 11/04/2016 or 2016/04/11). Given the expected size of the datasets, sets of blocking attributes will be selected (e.g., sex, date of birth, initials) and record pairs with the same matched attributes within blocks compared. After, record pairs will be compared for each linkage variable and an agreement score computed. This score will be used to weight the probability of a record pair belonging to the same child.

After obtaining the final database, person-time incidence rates for primary outcomes will be computed. Kaplan Meier method will be used to compare the probability of surviving 1st and 5th year of life or of not having a hospitalization, emergency department visit, a mild/ severe morbidity episode during the follow-up period according to exposure. Log rank test will be used for differences in survival rates between exposed and non-exposed children and hazard ratios (with confidence intervals) for quantifying the differences. Proportional hazards regression analysis will be used to explore the effects of several variables on the survival outcomes. If missing data is below 5%, we will use complete-case analysis. Otherwise, the frequency and patterns of missing data will be analysed and if appropriate, multiple imputation techniques used.

Confounders to be measured (and controlled for) are sex, health unit, completeness of and timeliness of vaccination status and scheme, socioeconomic status and BCG strain.

ELIGIBILITY:
Inclusion Criteria:

* children born in Portugal, live-births and births coded as DRG 795 (normal new-born)

Exclusion Criteria:

* new-borns with low-birth weight (<2kg), premature (<37 weeks) and known or suspected HIV infection

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Under-5 children born and registered in Portugal between 1 July 2010 and 30 June 2021.
Sampling Method: Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | First 5 years of life or until 30 June 2022
  Person time incidence rate of death (all causes)
Mortality due to TB | First 5 years of life or until 30 June 2022
  Person time incidence rate of death (TB)
Mild morbidity | First 5 years of life or until 30 June 2022
  Contacts with the medical doctor or nurse at a primary health center unit due to disease or ill-health during the follow-up, besides contacts related to recommended child-surveillance scheme or other reasons besides health
Severe morbidity | First 5 years of life or until 30 June 2022
  Hospitalization and/or visits to the emergency department
TB | First 5 years of life or until 30 June 2022
  Confirmed case of TB

SECONDARY OUTCOMES:
Mortality profile of under-5 children between 2010 and 2022 | 2010 to 2022
  Description of causes of death, time, sex and age distribution
Morbidity profile of under-5 children between 2010 and 2022 | 2010 to 2022
  Main causes of ill-health that required visit to health services (primary and emergency department) or hospitalization, time, sex and age distribution
Profile of non-vaccinated children before and after 2016 | 2010 to 2022
  Socio-demographic and clinical characteristics of children who did not received BCG
NHS hospital and PHC utilization profile of under-5 children | 2010 to 2022
  Main causes for seeking health care in PHC and in hospitals, time, age, sex distribution, clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Ines Fronteira, PhD, Principal Investigator — Instituto de Higiene e Medicina Tropical - Universidade Nova de Lisboa
Locations (1):
- Instituto de Higiene e Medicina Tropical, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fronteira I, Pacheco M, Schaltz-Buchholzer F, Ferrinho P. Nonspecific Effects of the Bacillus Calmette-Guerin Vaccine in Portuguese Children Under 5 Years of Age: Protocol for a Population-Based Historical Birth Cohort Study. JMIR Res Protoc. 2024 Mar 14;13:e55332. doi: 10.2196/55332. PMID 38328938